CLINICAL TRIAL: NCT00334568
Title: A Double-blind, Randomised, Placebo-controlled, Parallel-group Study to Investigate the Effects of Rosiglitazone (Extended Release Tablets) on Cerebral Glucose Utilisation and Cognition in Subjects With Mild to Moderate Alzheimers Disease (AD)
Brief Title: Effects Of Rosiglitazone (Extended Release Tablets) On Cerebral Glucose Utilisation And Cognition Alzheimers Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVA100930
Record Dates: First submitted 2006-06-06; First posted 2006-06-08 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Alzheimer's Disease
Keywords: AVANDIA; Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Rosi XR (Experimental): Rosi XR
  Interventions: Drug: Rosiglitazone XR (extended release) oral tablets
- Placebo (Placebo Comparator): Placebo (matched)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone XR (extended release) oral tablets — Rosi XR tablets
  Arms: Rosi XR
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Clinical features in patients with the familial early onset forms and the sporadic forms of Alzheimers disease are similar, although the course of deterioration may be different. It would be very informative to examine the drug response of patients with Alzheimers disease by a certain genotype to find evidence favouring genotype-specific drug responses that may indicate genetically defined phenotypic differences in alzheimers disease.

ELIGIBILITY:
Inclusion Criteria:

* Meets the National Institute of Neurological and Communicative Diseases and Stroke/Alzheimers Disease and Related Disorders Association (NINCDS-ADRDA) criteria for Alzheimers disease, regardless of date of diagnosis relative to study entry date.
* Has an Alzheimers disease status of mild to moderate, as classified by a Mini Mental State Examination (MMSE) score of 16 - 26 inclusive at screening.
* Post-menopausal females defined as menopause is defined as >6 months without menstrual period with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms. However if indicated this should be confirmed by oestradiol and FSH levels consistent with menopause (according to local laboratory ranges).
* Women who are on HRT (hormone replacement therapy) treatment, and have not been confirmed as post-menopausal should be advised to use contraception.
* Has a permanent caregiver who is willing to attend all visits, oversee the subjects compliance with protocol-specified procedures and study medication, and report on subjects status. (Subjects living alone or in a nursing home are not eligible).

Exclusion Criteria:

* Has a history of or suffers from claustrophobia.
* Is unable to lie comfortably on a bed inside a PET camera with their head in the field of view for at least 60 minutes as assessed by physical examination and medical history (e.g. back pain, arthritis).
* Has a history or presence of other neurological or other medical conditions that may influence the outcome or analysis of the PET scan results. Examples of such conditions include, but are not limited to stroke, traumatic brain injury, epilepsy or space occupying lesions.
* History of Type I or Type II diabetes mellitus.
* Fasting plasma glucose level >126 mg/dL (>7.0 mmol/L) or HbA1c >6.2%.
* History or clinical/laboratory evidence of moderate congestive heart failure defined by the New York Heart Association criteria (class II-IV.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in global and regional cerebral glucose metabolism/Cerebral Metabolic Rate for glucose (CMRglu) as measured by the ratio of Ki to K1 | at baseline and 12 months.

SECONDARY OUTCOMES:
Changes in global and regional CMRglu as measured by [18F]FDG uptake. | between baseline and 12 month point
Global changes in brain structure from baseline as measured by structural MRI from baseline.Vital signs and ECGs. | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom